CLINICAL TRIAL: NCT00217711
Title: Oxaliplatin, Irinotecan, and Capecitabine as a Combination Regimen for First-Line Treatment of Advanced or Metastatic Colorectal Cancer
Brief Title: Oxaliplatin, Irinotecan, and Capecitabine in Treating Patients With Advanced or Metastatic Colorectal Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/03; EU-20524
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Irinotecan; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Active Comparator): Oxaliplatin, Irinotecan, and Capecitabine
  Interventions: Drug: Capecitabine; Drug: irinotecan hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — capecitabine
Drug: irinotecan hydrochloride — irinotecan hydrochloride
Drug: oxaliplatin — oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, irinotecan, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of capecitabine when given together with oxaliplatin and irinotecan and to see how well they work in treating patients with advanced or metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of capecitabine administered in combination with oxaliplatin and irinotecan in patients with unresectable advanced or metastatic colorectal cancer. (Phase I)
* Determine the efficacy of this regimen in these patients. (Phase II)

Secondary

* Determine the tolerability of this regimen in these patients. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study of capecitabine followed by a phase II study.

* Phase I: Patients receive oxaliplatin IV over 2 hours on days 1 and 15, irinotecan IV over 1 hour on days 8 and 22, and oral capecitabine twice daily on days 1-29. Treatment repeats every 5 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive capecitabine at the MTD and irinotecan and oxaliplatin as in phase I.

After completion of study treatment, patients are followed every 2 months for 1 year and then every 4 months thereafter.

PROJECTED ACCRUAL: A total of 23-32 patients (3-12 for the phase I portion and 20 for the phase II portion) will be accrued for this study within 2.75 years

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable advanced or metastatic colorectal cancer
* Measurable disease (phase II only)

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan or MRI
* No presence or history of CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.25 times upper limit of normal (ULN) (1.5 times ULN if liver metastases are present)
* AST and ALT ≤ 3 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine clearance > 60 mL/min

Cardiovascular

* No New York Heart Association class III-IV congestive heart failure
* No symptomatic coronary artery disease
* No uncontrolled cardiac arrhythmia
* No myocardial infarction within the past year
* No other clinically significant cardiac disease

Immunologic

* No active autoimmune disease
* No uncontrolled infection
* No prior severe reaction to fluoropyrimidine therapy or known hypersensitivity to fluorouracil
* No known hypersensitivity to any component of study drugs

Other

* Not pregnant or nursing
* Negative pregnancy test
* Patients must use effective contraception during and for 1 year after study participation
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No peripheral neuropathy > grade 1 of any origin (e.g., alcohol or diabetes)
* No nausea, vomiting, or malabsorption syndrome that would preclude ingestion or absorption of oral medication
* No psychiatric disability that would preclude study compliance
* No uncontrolled diabetes
* No other serious underlying medical condition that would preclude study participation
* No known dihydropyrimidine dehydrogenase deficiency

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic hematopoietic growth factors

Chemotherapy

* More than 6 months since prior adjuvant fluoropyrimidine chemotherapy
* No other prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy

  * Concurrent radiotherapy of a single painful lesion allowed

Surgery

* Not specified

Other

* More than 30 days since prior clinical trial participation
* No other concurrent experimental drugs
* No other concurrent anticancer therapy
* No concurrent sorivudine or its chemically-related analogues (e.g., lamivudine)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
capecitabine + oxaliplatin + irinotecan dose finding | 30 days
  Determine the maximum tolerated dose and recommended phase II dose of capecitabine administered in combination with oxaliplatin and irinotecan in patients with unresectable advanced or metastatic colorectal cancer. (Phase I)
Efficacy of Oxaliplatin, Irinotecan, and Capecitabine | 2 months
  Determine the efficacy of this regimen in these patients (Phase II)

SECONDARY OUTCOMES:
Objective response (CR or PR) as measured after completion of study treatment | 2 months
Adverse events as measured after completion of study treatment | 2 months
Time to progression | life-long
Time to treatment failure as measured after completion of study treatment | life-long
Overall survival | life-long

CONTACTS AND LOCATIONS:
Overall Officials: Razvan Popescu, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (4):
- Switzerland (4):
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Hirslanden Klinik Aarau, Lausanne
  - City Hospital Triemli, Zurich

REFERENCES:
- [Result] von Moos R, Roth A, Ruhstaller T, Widmer L, Uhlmann C, Cathomas R, Koberle D, Simcock M, Lanz D, Popescu R. Oxaliplatin, irinotecan and capecitabine (OCX) for first-line treatment of advanced/metastatic colorectal cancer: a phase I trial (SAKK 41/03). Onkologie. 2010;33(6):295-9. doi: 10.1159/000313598. Epub 2010 May 14. PMID 20523092